CLINICAL TRIAL: NCT05321134
Title: Evaluation of SINGLE PORT (SP) Robotic Technology in Colorectal Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: University of California, San Francisco (Other); Yale University (Other); Henry Ford Hospital (Other); University of Massachusetts, Worcester (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022178
Record Dates: First submitted 2022-03-31; First posted 2022-04-11 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Colo-rectal Cancer; Rectal Prolapse; Colostomy Stoma; Colorectal Disorders
Keywords: robotic surgery; colorectal surgery; single port; Intuitive SP platform
MeSH Terms: conditions — Colonic Neoplasms; Rectal Prolapse

STUDY DESIGN:
Intervention Model Description: Single center, prospective, open-label, investigator initiated, non-randomized, interventional case-control study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Single Port Robotic Surgery Arm (Experimental): Study subjects will undergo the colorectal surgical procedure (determined based on routine standard clinical care) using the Intuitive Da Vinci Single Port SP system
  Interventions: Device: Single port robotic colorectal surgical procedure

INTERVENTIONS:
Device: Single port robotic colorectal surgical procedure — After screening and counseling, study subjects who wish to participate will undergo the colorectal surgical procedure (determined based on routine standard clinical care) using the alternate Intuitive Da Vinci Single Port SP system rather than the currently used multiport system, (Intuitive Da Vinci Multiport Xi System).
  Using standardized case report forms, the investigators will track clinical parameters and describe the safety & quality event rate for SP platform transabdominal and transanal colorectal operations.

SUMMARY:
Currently a multiport robotic surgery platform (Intuitive Xi) is widely available and used for colorectal surgery indications. A Single port platform (Intuitive SP) is FDA approved for Head and Neck and Urology but has not been widely used in colorectal surgery. This study seeks to evaluate the safe and effective use of the SP platform for colorectal surgery indications.

DETAILED DESCRIPTION:
This is a single center, prospective, open-label, investigator initiated, non-randomized, interventional case-control study where researchers will study colorectal surgical procedures done using the novel Single Port (SP) Robotic Platform and compare perioperative outcomes to colorectal surgical cases done using the traditional Multi-port (Xi) Robotic Platform.

AIM 1 To assess the feasibility and safety/quality of a SP platform for transabdominal and transanal colorectal operations which are currently done using multiport robotic platforms.

AIM 2 To evaluate safety and quality outcomes post SP surgery in comparison with contemporaneous standard multiport Xi platform procedures.

ELIGIBILITY:
Inclusion Criteria:

* The subject is male or female, greater than or equal to 18 years of age. If female, the subject has a negative urine pregnancy test and is not lactating, or has not been of childbearing potential for at least 3 months prior to use of study product. To be considered to be not of childbearing potential, the subject must be postmenopausal for at least 2 years; have had a hysterectomy or bilateral tubal ligation, or be proven to be otherwise incapable of pregnancy. If of childbearing potential, the subject must have been practicing one of the following methods of contraception consistently for at least 1 month prior to study entry and agree to continue practicing it during the study: hormonal contraceptives, intrauterine device, spermicide and barrier, spouse/partner sterility; or is practicing abstinence and agrees to continue abstinence or to start an acceptable method of contraception from the above list if sexual activity commences.
* There is documentation of a colorectal diagnosis requiring operative interventions with clinical plans for a robotic operation.
* For robotic transanal procedures, patients who would meet standard guidelines for a transanal procedures (T1N0 rectal adenocarcinoma, Precancerous adenomas, and localized neuroendocrine tumors) distal to 15 cm from the anal verge.
* The subject is in good general health as evidenced by medical history and physical examination
* The subject is able and willing to provide written informed consent.
* The subject agrees to comply with the requirements of the protocol and complete study measures.
* The subject has stable residence and telephone.

Exclusion Criteria:

* The subject is child less than 18 years of age
* The subject is a female who is pregnant or lactating
* The subject falls under the American Society of Anesthesia Class IV (Patients with severe systemic disease that is a constant threat to life).
* The subject falls under American Society of Anesthesia Class V (Moribund patients who is not expected to survive without the operation)
* The subject has a history of clinically significant renal, hepatic, neurological, cardiac or chronic pulmonary disease that in the judgment of the investigator precludes participation.
* The subject has advanced/ Stage IV cancer
* The subject has received neo-adjuvant chemotherapy or radiation therapy
* The subject requires an emergency operation.
* The subject is unable to fully comprehend or consent to the study
* The subject is unwilling to be available for follow-up assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-04-28 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Assess safety & quality event rate for SP platform transabdominal and transanal colorectal operations | 30 days
  A safety & quality event will be defined as occurring if any of the following occur:
  * Conversion to open or laparoscopic procedure
  * EBL > 200 ml, or
  * Operative time > 90th percentile of all procedures with matching CPT code, or
  * Positive pathological margins (if applicable), or
  * Fragmented specimen (if applicable) or
  * Unplanned ICU stay or
  * Post-procedure LOS > 90th percentile of all procedures with matching CPT code, or
  * Reoperation within 30 days or
  * Post Procedure Pain > 90th percentile (visual analog score)
  * Postoperative complication as defined by NSQIP (including SSI, DVT, PE, readmission, anastomotic Leak (if applicable)

CONTACTS AND LOCATIONS:
Overall Officials: Ankit Sarin, MD, Principal Investigator — University of California, Davis
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sarin A, Barnes KE, Shui AM, Nakamura Y, Hoffman DB, Romero-Hernandez F, Chern H. Initial Experience With Single-Port Robotic Right Colectomies: Results of an Investigator-Initiated Investigational Device Exemption Study Using a Novel Single-Port Robotic Platform. Dis Colon Rectum. 2024 Oct 1;67(10):e1600-e1606. doi: 10.1097/DCR.0000000000003352. Epub 2024 Sep 5. PMID 39250792